CLINICAL TRIAL: NCT06576544
Title: Evidence-Based Prediction and Prevention of Adverse Outcomes Caused by Postpartum Hypertension
Brief Title: Wearables to Define Postpartum Blood Pressure Trajectories and Facilitate Evidence-based Monitoring Guidelines
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ukachi Emeruwa, Assistant Professor, University of California, San Diego
Other Study IDs: 808180
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Hypertension, Pregnancy-Induced; Hypertension; Postpartum Preeclampsia; Postpartum Complication; Postpartum Pre-Eclampsia; Cardiovascular Diseases; Cardiovascular Morbidity; Morbidity;Perinatal
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-risk: Individuals having chronic HTN, according to ACOG guidelines, as either SBP ≥140 mmHg or DBP ≥90 mmHg on at least 2 occasions, ≥4 hours apart, prior to 20 weeks gestation
  Interventions: Device: BP Watch
- Intermediate-risk: Individuals who are at risk of de novo PP HTN; these are individuals who are at risk for preeclampsia based on an adapted USPSTF algorithm but who did not develop HTN by the time of delivery. The algorithm is as follows:
  -One or more of the following high risk conditions and/or two or more of the following moderate risk conditions for development of de novo postpartum hypertension: i. High risk conditions: pregestational diabetes mellitus, renal disease, autoimmune disease (systemic lupus erythematosus, antiphospholipid syndrome), multifetal gestation, gestational diabetes mellitus A2 (i.e. medication-dependent), history of preeclampsia in a prior pregnancy (not including the index pregnancy) ii. Moderate risk conditions: primiparity, obesity (BMI ≥ 35 kg/m2), age ≥ 35 years, Black or African-American race, family history of preeclampsia
  Interventions: Device: BP Watch
- Low-risk: Having no diagnosis of HTN/HDP by the time of delivery and not meeting criteria for increased risk of HDP or de novo PP HTN.
  Interventions: Device: BP Watch

INTERVENTIONS:
Device: BP Watch — Participants are given a non-invasive wearable device that monitors blood pressure multiple times daily for 6 weeks postpartum.

SUMMARY:
To better understand postpartum blood pressure changes, the investigators are proposing a study to monitor blood pressure after delivery in 100 patients who the investigators expect to have normal blood pressure (i.e. low-risk group), 100 patients who the investigators expect to be at risk of new-onset high blood pressure postpartum (i.e. intermediate-risk group), and 100 patients who had high blood pressure prior to pregnancy (or very early, before 20 weeks in pregnancy) who the investigators know are at high risk of blood-pressure related complications postpartum (i.e. high-risk group). Patients will be given a non-invasive wearable device that monitors blood pressure continuously for 6 weeks postpartum. The investigators expect that the daily changes in blood pressure will be different between these groups, which may allow us to better predict who is at risk, how much monitoring is needed, and when to intervene before the blood pressure abnormalities cause complications. The blood pressure device that will be given to patients is the YHE® BP Doctor Med Blood Pressure Smartwatch. This is a highly-accurate medical grade device that has not received FDA clearance. As such, the device is not being used to make blood pressure management and treatment decisions, but rather to gather data on postpartum cardiovascular physiology. Safety stops are built into the protocol such that elevated readings detected by the watch will trigger clinical referrals and validation by standard blood pressure cuffs prior to determine need for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum birthing person 18 years of age or older
* At least 20 weeks gestation at time of delivery
* Meeting criteria for 1 of 3 risk categories for PP HTN and hypertensive morbidity
* Planned postpartum care at UCSD

Exclusion Criteria:

* Inability to give informed consent
* Institutionalization for psychiatric disorder, mental deficiency or incarcerated
* Initiation of antihypertensive therapy prior to discharge from delivery hospitalization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The present research study focuses on postpartum hypertension. The target sample size is 300 postpartum patients delivering at UCSD. Within this population, we aim to enroll 100 low-risk participants, 100 intermediate-risk participants, and 100 high-risk participants.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postpartum blood pressure trends | 6 week postpartum period
  Define the differences in longitudinal trends in blood pressure during the 6-week postpartum period between (a) subjects at low-risk for postpartum hypertension, (b) an intermediate-risk group, and (c) those at high-risk for postpartum hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobs Medical Center at UC San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, IPD will be shared under controlled access
Supporting Information: Study Protocol
Time Frame: IPD will be shared once primary analysis is completed
Access Criteria: IPD will be shared under controlled access (e.g. Via DASH: https://catalog.data.gov/dataset/nih-data-and-specimen-hub-dash).
URL: https://catalog.data.gov/dataset/nih-data-and-specimen-hub-dash